CLINICAL TRIAL: NCT03029923
Title: Integrated Smoking Cessation and Mood Management for ACS Patients (PACES Phase IV Vanguard R56 Trial)
Brief Title: Integrated Smoking Cessation and Mood Management for ACS Patients
Acronym: PACES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for this pilot transitioned into funding for a fully powered study.
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Andrew Busch, Assistant Professor, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 214016; R56HL131711-01A1 (NIH)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Acute Coronary Syndrome; Tobacco Use
Keywords: smoking; depression; Behavioral Activation
MeSH Terms: conditions — Acute Coronary Syndrome; Tobacco Use; Smoking; Depression | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking Cessation and Mood Management (Experimental): Participants will receive standard smoking cessation plus Behavioral Activation based mood management. Will be offered the nicotine patch if medically cleared.
  Interventions: Behavioral: Experimental: Behavioral Activation Treatment for Cardiac Smokers (BAT-CS)
- Smoking cessation and Health and Wellness (Active Comparator): Participants will receive standard smoking cessation plus health and wellness education. Will be offered the nicotine patch if medically cleared.
  Interventions: Behavioral: Smoking cessation plus Health and Wellness

INTERVENTIONS:
Behavioral: Experimental: Behavioral Activation Treatment for Cardiac Smokers (BAT-CS) — All participants will receive one hour of standard smoking cessation counseling during their hospitalization for an acute coronary syndrome. Participants will be randomized 1 week after discharge. Those assigned to BAT-CS condition will receive 5 more counseling sessions over the 12 weeks after discharge. The first will be up to one hour and will be conducted in person. The next 4 sessions will occur by phone and will take about 30 minutes. Post-discharge sessions will be focused on smoking cessation and mood management using behavioral activation techniques. Participants will be offered the nicotine patch if medically cleared.
  Arms: Smoking Cessation and Mood Management
Behavioral: Smoking cessation plus Health and Wellness — All participants will receive one hour of standard smoking cessation counseling during their hospitalization for an acute coronary syndrome. Participants will be randomized 1 week after discharge. Those assigned to the Smoking cessation plus Health and Wellness condition will receive 5 more counseling sessions over the 12 weeks after hospital discharge. The first will be up to one hour and will be conducted in person. The next 4 sessions will occur over the phone and will take about 30 minutes. Post-discharge sessions will be focused on smoking cessation and didactic health and wellness education. Participants will be offered the nicotine patch if medically cleared.
  Arms: Smoking cessation and Health and Wellness

SUMMARY:
Quitting smoking following acute coronary syndrome can reduce mortality up to 50%. However, depression and smoking are highly co-morbid and depressed mood may interfere with cessation and independently predicts mortality. Thus, a single, integrated treatment for both smoking and depression could be highly effective in reducing post-acute coronary syndrome mortality. Behavioral Activation (BA) is a well established treatment for depression and has recently shown promise as a treatment for smoking cessation. The investigators systematically developed an intervention integrating gold standard smoking cessation counseling with existing BA based mood management techniques for post-ACS smokers; Behavioral Activation Treatment for Cardiac Smokers (BAT-CS).

Objective: For this R56 the investigators will conduct a vanguard trial to pilot all methods, materials, and systems for the later fully powered BAT-CS vs. attention control trial. The investigators will enroll up to 36 smokers with ACS and randomize them to 12 weeks of BAT-CS or an attention control (Health and Wellness Education). Both groups will be offered the nicotine patch if medically safe.

ELIGIBILITY:
Inclusion Criteria:

1. hospital inpatients with an ACS diagnosis documented in medical record,
2. smoked 1 or more cigarettes per day before being hospitalized,
3. age of 18-75,
4. English fluency,
5. lives within a 1 hour drive of the admitting hospital and has no plans to move away from the area for 1 year,
6. willing to consider quitting smoking at discharge,
7. has telephone, and
8. willing to consent to all study procedures.

Exclusion Criteria:

1. limited mental competency (i.e., Mini Mental Status Exam score ≤ 23);
2. presence of severe mental illness that would interfere with participation (e.g., schizophrenia) or suicidality;
3. expected discharge to hospice; and
4. currently attending counseling for depression or smoking cessation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Estimated); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Acceptability | 12 weeks post-Discharge
  Treatment Acceptability as measured by the Client Satisfaction Questionnaire

SECONDARY OUTCOMES:
Smoking Cessation | 12 weeks post-Discharge
  7 day point-prevalence abstinence. Biochemically verified.
Depression Symptoms | 12 weeks post-Discharge
  Depression Symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9)

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No